CLINICAL TRIAL: NCT02884011
Title: Evaluating the Effect of Chronic Antihypertensive Therapy on Vasopressor Dosing in Septic Shock
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16081001
Record Dates: First submitted 2016-08-12; First posted 2016-08-30 (Estimated); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Septic Shock
Keywords: Chronic antihypertensives; Septic shock; Vasopressor; Vasopressor dosing
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- No chronic antihypertensives: not on either a chronic β-blocker or ACE-Inhibitor
- β-blocker: on chronic β-blocker
- ACE-Inhibitor: on chronic ACE-Inhibitor
- Both β-blocker and ACE-inhibitor: on both chronic β-blocker and ACE-inhibitor

SUMMARY:
Retrospective study to examine the effects of chronic antihypertensive medications on vasopressor dosing in septic shock

DETAILED DESCRIPTION:
This will be a retrospective four-cohort study. The four cohorts will be septic shock patients that were: 1) not on either a chronic β-blocker or chronic angiotensin-converting-enzyme inhibitor (ACE-Inhibitor), 2) on chronic β-blocker, 3) on ACE-Inhibitor, and 4) on both chronic β-blocker and ACE-inhibitor

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older
* Diagnosis of septic shock requiring vasopressor therapy (norepinephrine, epinephrine, phenylephrine, dopamine, or vasopressin)
* Admitted to an intensive care unit (ICU) at Rush University Medical Center (RUMC)
* Time frame: 01/01/2012 to 07/1/2016

Exclusion Criteria:

* Pregnant patients
* Transfer from outside hospital on vasopressors
* Admitted in cardiopulmonary arrest
* Prior arrest within 24 hours of admission to RUMC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, non-pregnant medical intensive care unite (MICU) patients with septic shock requiring vasopressor support
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua DeMott, Pharm.D., Principal Investigator — Rush University Medical Center; Ishaq Lat, Pharm.D., Principal Investigator — Rush University Medical Center; Gourang Patel, Pharm.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush Univeristy Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: retrospective study
Period: Overall Study
Arm/Group | No Chronic Antihypertensives | β-blocker | ACE-Inhibitor | Both β-blocker and ACE-inhibitor
Started | 51 | 46 | 17 | 19
Completed | 51 | 46 | 17 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Chronic Antihypertensives | β-blocker | ACE-Inhibitor | Both β-blocker and ACE-inhibitor | Total
Number analyzed (Participants) | 51 | 46 | 17 | 19 | 133
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [51 to 73] | 67 [57 to 72] | 70 [57 to 77] | 66 [62 to 73] | 65 [52 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 7 | 11 | 59
  Male | 32 | 24 | 10 | 8 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 18 | 27 | 6 | 9 | 60
  White | 23 | 15 | 8 | 7 | 53
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 4 | 3 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Total Vasopressor Dose
Description: The primary objective is to determine the effect of chronic β-blocker or ACE-inhibitor on vasopressor dosing in the first 48 hours of septic shock. Vasopressor types and cumulative doses including: norepinephrine, epinephrine, phenylephrine, dopamine, and vasopressin. Epinephrine, phenylephrine, and dopamine will be converted to norepinephrine equivalents in concordance with other literature: 100 mcg dopamine equivalent to 1 mcg norepinephrine, 1 mcg epinephrine equivalent to 1 mcg norepinephrine, and 2.2 mcg phenylephrine equivalent to 1 mcg norepinephrine
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: mg
Groups:
- No Beta-blocker or ACE Inhibitor: No beta-blocker or ACE inhibitor
- Beta-blocker Only: Beta-blocker only
- Ace Inhibitor: Ace inhibitor
- Beta-blocker and ACE Inhibitor: Beta-blocker and ACE inhibitor
Arm/Group | No Beta-blocker or ACE Inhibitor | Beta-blocker Only | Ace Inhibitor | Beta-blocker and ACE Inhibitor
Number analyzed (Participants) | 51 | 46 | 17 | 19
mg | 13.7 [6.0 to 35.7] | 13.1 [5.4 to 23.9] | 13.2 [1.2 to 36.7] | 11.3 [4.7 to 42.9]

2. Secondary Outcome: 30 mL/kg Fluid Within 6h
Description: Number of Participants with 30 mL/kg Fluid Within 6 Hours
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Groups:
- No Beta-blocker or ACE Inhibitor: Septic shock patients that were not on either a chronic β-blocker or chronic angiotensin-converting-enzyme inhibitor (ACE-Inhibitor)
- Beta-blocker Only: Septic shock patients that were on chronic β-blocker.
- Ace Inhibitor: Septic shock patients that were on ACE-Inhibitor.
- Beta-blocker and ACE Inhibitor: Septic shock patients that were on both chronic β-blocker and ACE-inhibitor.
Arm/Group | No Beta-blocker or ACE Inhibitor | Beta-blocker Only | Ace Inhibitor | Beta-blocker and ACE Inhibitor
Number analyzed (Participants) | 51 | 46 | 17 | 19
Participants | 36 | 27 | 12 | 16

3. Secondary Outcome: Inotrope Use
Description: Cumulative inotrope use at different time points (total mg). Example inotropes include dobutamine and milrinone
Time Frame: 6, 12, 24, 48 hours
Reporting Status: Not Posted

4. Secondary Outcome: Hydrocortisone Use
Description: Cumulative hydrocortisone (mg) use at different time points
Time Frame: 6, 12, 24, 48 hours
Reporting Status: Not Posted

5. Secondary Outcome: Cumulative Vasopressor Dose for Patients Receiving Other Antihypertensives
Description: To determine cumulative vasopressor dose at various time points of patients on chronic calcium channel blocker or other antihypertensives (i.e., hydralazine, clonidine, angiotensin-receptor-blocker (ARB), etc). Vasopressor types and cumulative doses including: norepinephrine, epinephrine, phenylephrine, dopamine, and vasopressin. Epinephrine, phenylephrine, and dopamine will be converted to norepinephrine equivalents in concordance with other literature: 100 mcg dopamine equivalent to 1 mcg norepinephrine, 1 mcg epinephrine equivalent to 1 mcg norepinephrine, and 2.2 mcg phenylephrine equivalent to 1 mcg norepinephrine
Time Frame: 6, 12, 24, 48 hours
Reporting Status: Not Posted

6. Secondary Outcome: 6-hour Vasopressor Dose
Description: Vasopressor types and cumulative doses including: norepinephrine, epinephrine, phenylephrine, dopamine, and vasopressin. Epinephrine, phenylephrine, and dopamine will be converted to norepinephrine equivalents in concordance with other literature: 100 mcg dopamine equivalent to 1 mcg norepinephrine, 1 mcg epinephrine equivalent to 1 mcg norepinephrine, and 2.2 mcg phenylephrine equivalent to 1 mcg norepinephrine
Time Frame: 6 hours
Reporting Status: Not Posted

7. Secondary Outcome: 12-hour Vasopressor Dose
Description: as for outcome 6
Time Frame: 12 hours
Reporting Status: Not Posted

8. Secondary Outcome: 24-hour Vasopressor Dose
Description: as for outcome 6
Time Frame: 24 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During the inpatient hospital stay, up to 48 hours
Description: inpatient mortality
Arm/Group | No Chronic Antihypertensives | β-blocker | ACE-Inhibitor | Both β-blocker and ACE-inhibitor
All-Cause Mortality (participants affected / at risk) | 21/51 | 26/46 | 6/17 | 11/19
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/46 | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/51 | 0/46 | 0/17 | 0/19

LIMITATIONS AND CAVEATS:
Adherence to prescribed chronic β-blockers or ACE inhibitors could not be confirmed. The electronic medical record charting by the staff may be subject to inaccuracies in vasopressor dose infusion changes and documentation. Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT02884011/Prot_SAP_000.pdf